CLINICAL TRIAL: NCT04974957
Title: A Multicenter, Open-Label, Phase Ib/II Trial of SHR-1701 Plus BP102 in Subjects With Selected Solid Tumors
Brief Title: Study of SHR-1701 Plus BP102 in Subjects With Selected Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701-II-207-LC
Record Dates: First submitted 2021-07-16; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1701+BP102 (Experimental)
  Interventions: Drug: SHR-1701；BP102

INTERVENTIONS:
Drug: SHR-1701；BP102 — Drug: SHR-1701 IV infusion
  Drug: BP102 IV infusion

SUMMARY:
The main purpose of this study was to assess the safety,efficacy and pharmacokinetic when combining SHR-1701 and BP102 in participants with advanced or metastatic non-squamous non-small cell lung cancer. To explore the immunogenicity of SHR-1701 and the relationship between corresponding biomarkers and therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced or metastatic non-squamous non-small cell lung cancer.
2. Failed with prior systemic treatments.
3. Measurable disease, as defined by RECIST v1.1
4. The Eastern Cancer Cooperative Group (ECOG) performance status of 0 or 1
5. Life expectancy ≥ 3 months
6. Adequate hematologic and end-organ function as defined in the protocol

Exclusion Criteria:

1. Histologically or cytologically confirmed mixed SCLC and NSCLC.
2. Symptomatic, untreated or active central nervous system metastases.
3. Systemic therapy with immunosuppressive agents within 2 weeks prior to initiation of study treatment
4. With any active autoimmune disease or history of autoimmune disease.
5. Inadequately controlled hypertension.
6. Tumor infiltration into the great vessels on imaging.
7. History of hemoptysis ≥2.5ml per episode within 1 month prior to initiation of study treatment.
8. Uncontrolled tumor-related pain.
9. Patients with active hepatitis B or hepatitis C
10. Severe infections within 4 weeks prior to initiation of study treatment.
11. Active tuberculosis within one year prior to initiation of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2021-08-30 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
Disease control rate (DCR) | 2 years
Duration of response (DOR) | 2 years
Overall survival (OS) | 2 years